CLINICAL TRIAL: NCT05330091
Title: Garden of Life Once Daily Women's Probiotic: Vaginal pH and Quality of Life Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Garden of Life, LLC (Industry)
Collaborators: Validcare, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: VCODWP1
Record Dates: First submitted 2022-03-25; First posted 2022-04-15 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Vaginal Health
Keywords: Probiotics; Bacterial Vaginosis; Vaginal pH
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Women: Once Daily Women's Probiotic Placebo
  Interventions: Dietary Supplement: Once Daily Women's Probiotic; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Once Daily Women's Probiotic — Active product
Other: Placebo — Placebo product

SUMMARY:
This decentralized observational study is designed to understand the effects of daily consumption of once daily woman's probiotic (ODWP) on vaginal pH levels in healthy female populations ages 19-70 years of age across the United States.

DETAILED DESCRIPTION:
This decentralized observational study is designed to understand the effects of daily consumption of once daily woman's probiotic (ODWP) on vaginal pH levels in healthy female populations ages 19-70 years of age across the United States. Participants will be divided into two cohorts of 100 participants each; one with a history of vaginal bacteriosis and one with no history of bacterial vaginosis, with between 20-30 percent of the total participants being post-menopausal. Participants will be provided and trained to use pH tests on a daily basis over the course of four menstrual cycles (or equivalent time for amenorrheic participants). During the first cycle (or equivalent timeframe) of measurement, participants will not consume neither placebo or once daily woman's probiotics (ODWP); allowing the establishment of a baseline or wash out period prior to active consumption and measurement of effect.

Participants will receive ODWP at no charge for consumption over the course of the study. Participants will be instructed to start and continue consumption over three menstrual cycles (or equivalent timeframe) based on participant's menstrual status and her demonstrated ability to self-measure and report vaginal pH via the Validcare Study app based platform (aka "the app), which is provided as a free, downloadable 21 CFR Part 11 compliant interface for all patient facing activities and communication with/from the principal investigator for the study duration.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 19-70 (21-70 for residents of Mississippi)
2. Non-menopausal women must have a regular menstrual cycle (26-32 days)
3. Using birth control
4. Sexually active (intercourse at least 2x/month)
5. Agree to not introduce any other probiotic during the three months of study

Exclusion Criteria:

1. OCP or systemic hormonal contraception
2. No antibiotic treatment for at least 30 days
3. No active vaginal infection or symptoms of infection
4. No probiotic use for 30 days
5. Routine douching (except for immediately after menses)

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Health female population
Study Population: The population for this study will be generally healthy adults (19-70 years old) willing to consume ODWP or placebo of whom half have a history of bacterial vaginosis, and half who do not have such a history. Between 20-30% of the total population will be post- menopausal and will be distributed relatively equally between the 4 groups in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal pH | 4 months
  To compare the change in vaginal pH in both normal women and in normal women with a history of BV to and after treatment with Once Daily Women's Probiotic vs. placebo. Subjects will measure vaginal pH using a self-administered vaginal pH kit.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kaufmann, MD, Study Director — Validcare, LLC
Locations (1):
- Syzygy Research Solutions, Wellington, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with other researchers